CLINICAL TRIAL: NCT06073275
Title: Effects of Acute Beetroot Juice Intake on Performance, Maximal Oxygen Uptake, and Ventilatory Efficiency in Well-trained Master Rowers: A Randomized, Double-blinded Crossover Study
Brief Title: Effects of Beetroot Juice Intake on Performance and Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus docent Sant Joan de Déu-Universitat de Barcelona (Other)
Responsible Party: Principal Investigator, Manuel Vicente Garnacho Castano, Principal investigator, Campus docent Sant Joan de Déu-Universitat de Barcelona
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CDSJD
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Function; Nutrition, Healthy
Keywords: Cardiorespiratory performance; Time trial performance; Beetroot juice; Master rowers; well-trained

STUDY DESIGN:
Intervention Model Description: This study was a randomized, double-blind, crossover design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice intake (Experimental): Beetroot juice was administered 3 h before the start of the rowing ergometer test since the peak of nitrite in the blood occurs 2-3 h after nitrate ingestion. Beetroot juice was provided in a 140 mL maroon plastic bottle with no label. Participants were provided with a randomized bottle containing 140 mL (~12.8 mmol, ~808 mg of nitrate) of BRJ Beet-It-Pro Elite Shot concentrate (Beet IT; James White Drinks Ltd., Ipswich, UK).
  Interventions: Dietary Supplement: Beetroot juice ingestion
- Placebo intake (Placebo Comparator): Placebo was administered 3 h before the start of the rowing ergometer test. Placebo was provided in a 140 mL maroon plastic bottle with no label. Participants were provided with a randomized bottle containing 140 mL. The placebo drink was made by dissolving in 1 liter of water 2g of powdered SUPER BEETROOT (~ 0.01 mmol, 0.620 mg of nitrate, diet, food, Poland), 100% natural beetroot juice and organic label, and adding lemon juice to imitate the flavor and texture of the beetroot juice drink
  Interventions: Dietary Supplement: Placebo ingestion

INTERVENTIONS:
Dietary Supplement: Beetroot juice ingestion — Beetroot juice ingestion was randomly administered 3 h before the start of the test to the participants in two assessment sessions with a one-week washout between both sessions.
  Arms: Beetroot juice intake
Dietary Supplement: Placebo ingestion — Placebo ingestion was randomly administered 3 h before the start of the test to the participants in two assessment sessions with a one-week washout between both sessions.
  Arms: Placebo intake

SUMMARY:
This study was a randomized, double-blind, crossover design for 3 weeks. In the first week, a researcher explained all the experimental procedures to the participants. In the following two weeks, the participants attended the Exercise Physiology laboratory to be assessed in 2 rowing ergometer sessions, separated from each other by a washout period of 7 days, under the same environmental conditions.

In both strictly identical sessions, the participants randomly ingested beetroot juice (BRJ) or placebo (PL) 3 hours before the start of the tests.

DETAILED DESCRIPTION:
Three hours after BRJ or PL intake, the participants began the 2,000-meter rowing ergometer test. Before starting (pretest) and at the end of the tests (posttest), blood oxygen saturation, rating of perceived exertion (RPE), and blood lactate measurements were taken. During the rowing ergometer tests, performance parameters and cardiorespiratory variables were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. national and/or international level;
2. without cardiovascular, respiratory, metabolic, neurological or orthopedic disorders that may affect the performance of the rowing ergometer test;
3. no consumption of drugs or medicines;
4. no smoking;
5. Informed consent to participate in the study signed by all rowers

Exclusion Criteria:

1. Ingestion of nutritional supplements taken in the three months prior to the start of the study;
2. no following the guidelines established by the nutrition professional.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — well-trained male master rowers
Enrollment: 10 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Rowing performance: Time trial | through study completion, an average of 3 weeks
  minutes:seconds (mm:ss)
Rowing performance: Mean Power output | through study completion, an average of 3 weeks
  Watts
Rowing performance: meter per stroke | through study completion, an average of 3 weeks
  Meters
Cardiorespiratory performance: absolute oxygen uptake | through study completion, an average of 3 weeks
  V̇O2max (L/min)
Cardiorespiratory performance: relative oxygen uptake | through study completion, an average of 3 weeks
  V̇O2max (mL/kg/min)
Cardiorespiratory performance: ventilatory efficiency | through study completion, an average of 3 weeks
  slope of Ventilation/Carbon dioxide production
Metabolic performance: lactate | through study completion, an average of 3 weeks
  mmol/L

SECONDARY OUTCOMES:
Cardiorespiratory performance: Maximum heart rate | through study completion, an average of 3 weeks
  beats/min
Cardiorespiratory performance: Mean heart rate | through study completion, an average of 3 weeks
  beats/min
Saturation | through study completion, an average of 3 weeks
  percentage
Cardiorespiratory performance: minute ventilation | through study completion, an average of 3 weeks
  minute ventilation in L/min
Scale of Perceived exertion ratio (RPE) | through study completion, an average of 3 weeks
  Scale from 0 to 10. 0 = rest; 10 = maximum effort
Rowing performance: strokes | through study completion, an average of 3 weeks
  Mean strokes per minute

CONTACTS AND LOCATIONS:
Overall Officials: Manuel V Garnacho-Castaño, PhD, Principal Investigator — Campus docent Sant Joan de Déu-Universitat de Barcelona
Locations (1):
- Campus Docent Sant Joan de Déu. Universitat de Barcelona, Sant Boi de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No